CLINICAL TRIAL: NCT02249260
Title: Long-term Follow up of Exercise Based Cardiac Rehabilitation in Oslo
Brief Title: A Prospective Cohort Study of Heart Patients Included in Exercise Based Rehabilitation in Oslo
Acronym: OsloHeartEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Birgitta Blakstad Nilsson, PhD, Postdoc, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/553 (REK)
Record Dates: First submitted 2014-08-26; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Cardiac Disease
Keywords: Exercise, cardiac rehabilitation, quality of life
MeSH Terms: conditions — Heart Diseases; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral (Experimental): Group-based high intensity interval training and lifestyle counseling
  Interventions: Behavioral: High intensity interval training

INTERVENTIONS:
Behavioral: High intensity interval training — Group-based high-intensity aerobic interval training and lifestyle counseling
  Other Names: The Norwegian Ullevaal model

SUMMARY:
Outcomes evaluation is a critical component in outpatient cardiac rehabilitation. The aim of this study is to examine factors who predict long-term effects of improved peak oxygen uptake one year after participating in cardiac rehabilitation.

Secondary to evaluate the short and long-term outcome of a 12-week outpatient cardiac rehabilitation program.

DETAILED DESCRIPTION:
A prospective cohort study including all cardiac patients referred for outpatient cardiac rehabilitation in a primary care clinic in Oslo. The main efficacy variable is the changes in exercise capacity (VO2peak) as a primary prognostic measure of successful rehabilitation. HRQoL are measured by self-report using the COOP/WONCA questionnaire and SF-36.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary heart disease
* valvular surgery
* refered to high-intensity exercise training from a cardiologist

Exclusion Criteria:

* acute myocardial infarction within four week
* serious rhythm disturbances
* unstable angina pectoris
* known significant comorbidity
* symptomatic peripheral vascular disease
* obstructive pulmonary disease with forced expiratory vital capacity < 60% of predicted
* left ventricular ejection fraction < 40%

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen uptake | baseline, 15 months
  Change from baseline in peak oxygen uptake at 15 months

SECONDARY OUTCOMES:
Health related quality of life | baseline, 12 weeks
  Changes from baseline in quality of life (COOP/WONCA and SF-36) at 12 weeks
Peak oxygen uptake | baseline, 12 weeks
  Change from baseline in peak oxygen uptake at 12 weeks
Time to exhaustion | baseline, 15 months
  Change from baseline in "time to exhaustion" at 15 months
Time to exhaustion | baseline, 12 weeks
  Change from baseline in time to exhaustion at 12 weeks

OTHER OUTCOMES:
Systolic and diastolic Blood Pressure | baseline, 12 weeks
  Changes from baseline in systolic and diastolic blood pressure at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta B Nilsson, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Norwegian Sport Clinic (NIMI), Oslo, Oslo County, Norway